CLINICAL TRIAL: NCT05020496
Title: Role of Trem-1 in Ultraviolet Radiation-induced Immune Suppression
Brief Title: Trem-1 and Ultraviolet Radiation-induced Immune Suppression
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Nabiha Yusuf, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 300007159; R01 AI157398-01 (Other Grant/Funding Number: NIAID)
Record Dates: First submitted 2021-07-19; First posted 2021-08-25 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Skin Diseases
Keywords: immune suppression
MeSH Terms: conditions — Skin Diseases | interventions — diphenylcyclopropenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Negative Control, 20 participants) (No Intervention): At the first visit, various doses of diphenylcyclopropenone (DPCP) are applied in acetone to give the required dose range, increasing by 60% increments. Elicitation patch is applied on the upper inner arm skin and removed by patients themselves exactly 6 hours after the application.
  The second visit will be 48 hours after the DPCP treatment. At this visit, the bi-fold skin thickness will be measured using a Medical Skinfold Caliper.
  The group1 will have only one treatment with DPCP and serve as negative controls for DPCP induced cutaneous immune responses in comparison to Group 2 and 3, which require two treatments with DPCP (sensitization and challenge) as described in the following group 2 and 3. The first reading of skin thickness prior to DPCP application serves as the baseline and the second reading after DPCP indicates an increase in skin thickness, which represents a quantitative parameter of DPCP induced immune responses.
- Group 2 (Positive Control, 20 participants) (Other): This group of the study will take approximately 5 weeks and requires 3 visits. At the first visit, skin sites on the right upper buttock will be topically treated with a patch of the contact sensitizer (DPCP) for sensitization on the upper buttock for 48 hours. The skin patches will be removed by patients themselves after the application.
  The second visit will be four weeks after the DPCP sensitization, participants will have a DPCP treatment again on the right upper inner arm with the same agent. At the visit, the bi-fold skin thickness will be measured prior to the application of DPCP skin patch by using a Medical Skinfold Caliper. Various DPCP doses are applied increasing by 60% increments. The patches are applied on the upper inner arm skin and removed by patients themselves exactly 6 hours after application.
  The third and final visit will be 48 hours after the second DPCP treatment. At this visit, bi-fold skin thickness will be measured using a Caliper.
  Interventions: Drug: Diphenylcyclopropenone (DPCP)
- Group 3 (UVB & Biopsy 30 participants) (Experimental): This group of the study will take approximately 10 weeks and requires 10 visits.
  At the first visit, blood will be collected and MED will be determined. The second visit will be 24h after UV when MED will be measured. Blood will be collected from patients at this time. The third visit will be on the 8th day. The two marked skin sites will be UV exposed at 2MED on 4 consecutive days.
  Days 9-11 make up the fourth, fifth, and sixth visits. Following the last UV exposure blood will be collected. A single dose of DPCP will be placed on the upper buttock for 48 hours. The seventh visit will be on the 12th day when two skin biopsies will be taken. The ninth visit will be four weeks after the sensitization with DPCP, when the upper inner arm will be treated with DPCP. Bi-fold skin thickness will be measured prior to the application of DPCP. Various DPCP doses are applied. The tenth visit will be 48 hours after the DPCP treatment. At this visit, bi-fold skin thickness will be measured.
  Interventions: Drug: Diphenylcyclopropenone (DPCP)

INTERVENTIONS:
Drug: Diphenylcyclopropenone (DPCP) — Drug will be applied topically on the skin. It will cause contact hypersensitivity in patients
  Arms: Group 2 (Positive Control, 20 participants); Group 3 (UVB & Biopsy 30 participants)

SUMMARY:
The overall goal of this study is to determine novel mechanisms for ultraviolet light (UV)-induced suppression of the immune system in human subjects and to improve understanding of UV-induced skin carcinogenesis.

DETAILED DESCRIPTION:
Sunlight is the major environmental agent to which the skin is exposed. Injudicious exposure to wavelengths in the ultraviolet spectrum can lead to sunburn, aging of the skin, skin cancer and a variety of photosensitivity diseases, many of which have an immunologic pathogenesis. American Cancer Society acknowledges that most skin cancers are a direct result of exposure to the ultraviolet (UV) rays in sunlight. Skin cancer has also been linked to exposure to some artificial sources of UV rays (indoor tanning, welding and metal work, and phototherapy). UV, in addition to producing mutant cells, also impairs host cell-mediated immune responses that have evolved to identify and eradicate the mutant cells before they develop into clinically apparent malignancies. In fact, organ transplant recipients who are treated with immunosuppressive medications have a greatly increased risk (up to 100 times) of UV induced skin cancers and the tumors that do develop behave more aggressively. Triggering receptor expressed on myeloid cells (Trem)-1 is highly expressed by myeloid cells in human infectious and inflammatory diseases and is associated with poor prognosis of cancer patients. However, most studies have focused on Trem1 mediated effects on innate immune cells such as neutrophils in inflammatory reactions. Little is known about whether and how Trem1 regulates the adaptive immunity, especially the activity of antigen presenting cells (APC) to regulate the activation and function of antigen specific T cells. Our study will demonstrate a novel mechanism for Trem1 signaling in T cell mediated immune responses and photocarcinogenesis in skin. Different biological parameters in UV exposed skin tissues will be analyzed, which are crucial for UV-induced DNA damage, erythema, and immune suppressive effects that have been directly associated with photoimmunology and implicated in the risk of skin cancer. These will correlated with the responsiveness of allergen induced contact hypersensitivity.

Participants will be stratified based on gender and then randomly assigned to: 1) Control 2) Non-UVB, or 3) UVB groups. The primary endpoint for the study will be the CHS evaluation on day 34.The Control group no DPCP (Group 1) will serve as a negative control while the UVB & diphenylcyclopropenone (DPCP) group (Group 2) will serves as a positive control for measurement of response to irritant (contact hypersensitivity = CHS). Subjects in the UVB, DPCP, and Biopsy group (Group 3), who have no more than one standard deviation above the mean of CHS from the negative Control group, will be considered as Non-responders.

ELIGIBILITY:
* Inclusion Criteria
* Patient age 18-35
* Patient able to understand requirements of the study and risks involved
* Patient able to sign a consent form

Exclusion Criteria:

* Patients Fitzpatrick IV-VI
* A recent history of vitiligo, melasma, and other disorders of pigmentation with the exception of post inflammatory hyperpigmentation
* Patients with eczema, psoriasis, and contact dermatitis
* A known history of photosensitivity disorders
* A known history of melanoma or non-melanoma skin cancers
* Those planning on going to the tanning parlors
* Using any of the photosensitizing medication
* A woman who is lactating, pregnant, or planning to become pregnant
* Patient planning on exposing the irradiated or control areas to the sun
* Patients with organ transplantation, an immunodeficiency disorder or the use of an immunosuppressive drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Contact hypersensitivity | 24 hours after application
  Measurement of skin bifold thickness after application of DPCP in millimeter

CONTACTS AND LOCATIONS:
Overall Officials: Craig Elmets, MD, Study Director — Univ. of Alabama at Birmingham; Tyler Downing, MD, Study Director — University of Alabama at Birmingham
Locations (1):
- Whitaker Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No